CLINICAL TRIAL: NCT06772766
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of 9MW3011 in Patients With Non-transfusion-dependent β- Thalassemia
Brief Title: A Multiple Ascending Dose Study of 9MW3011 in Patients With Non-transfusion-dependent β-thalassemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 9MW3011-C04
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 9MW3011 or placebo (Randomized 4:1)
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- Cohort 2 (Experimental): 9MW3011 or placebo (Randomized 4:1)
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- Cohort 3 (Experimental): 9MW3011 or placebo (Randomized 4:1)
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- Cohort 4 (Experimental): 9MW3011 or placebo (Randomized 4:1)
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo

INTERVENTIONS:
Drug: 9MW3011 — Ascending IV doses administered per protocol
Drug: 9MW3011 placebo — Ascending IV doses administered per protocol

SUMMARY:
This is a phase Ib, randomized, double-blind, placebo-controlled, multiple ascending dose study . The objectives of the study are to evaluate the safety , tolerability, pharmacokinetics(PK), pharmacodynamics(PD), and immunogenicity of 9MW3011 in patients with non-transfusion-dependent β- thalassemia .

DETAILED DESCRIPTION:
A total of 40 subjects diagnosed with non-transfusion-dependent β-thalassemia will be enrolled in this study and assigned into four dosage cohorts. In each cohort, subjects will be randomized in a 4:1 ratio to receive 9MW3011 or placebo via intravenous infusion.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects aged 18 to 65 years (inclusive)
2. Subject must have a documented genetic diagnosis of β-thalassemia or hemoglobin E/ β-thalassemia
3. Subjects must meet the criteria for non-transfusion-dependent thalassemia
4. Subjects must have a baseline hemoglobin level between 70-100 g/L(inclusive), based on 2 consecutive measurements taken at least 1 week apart within 4 weeks before randomization
5. Subjects must have evidence of iron overload during screening
6. Subject must have performance status: Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
7. Subjects must fully understand the study procedures and methods, voluntarily participate in the trial, and sign an informed consent form

Key Exclusion Criteria:

1. Subjects diagnosed with alpha-thalassemia
2. Subjects diagnosed with HbS/beta-thalassemia or transfusion-dependent beta-thalassemia
3. Subjects exhibit severe iron overload at the time of screening
4. In addition to thalassemia, subjects have any other forms of anemia and hematological disorders that the investigator assesses may compromise safety or influence study outcomes
5. Combined with any significant systemic diseases or psychiatric disorders
6. Subjects have New York Heart Association (NYHA) Class III-IV heart failure and other cardiovascular diseases within 6 months prior to screening or currently present
7. During the screening or baseline period, subjects exhibiting a QTcF interval of ≥450ms for males and ≥470ms for females on a 12-lead electrocardiogram (ECG), or presenting an abnormal 12-lead ECG with clinical significance
8. Uncontrolled hypertension before screening
9. A history of malignant neoplasm occurring within the last five years
10. Severe infection requiring hospitalization or intravenous antimicrobial therapy, or uncontrolled systemic bacterial, fungal, or viral active infection
11. Subject have received concomitant treatment that was not permitted by the protocol
12. Subjects whose hematological parameters did not meet the inclusion criteria during screening
13. Subjects with a history of substance abuse, as well as those who yield positive results on substance abuse screening
14. Subjects who are unable to undergo MRI scans
15. Pregnant or lactating women
16. Subjects presenting any other factors deemed unsuitable for participation assessed by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(including serious adverse event) | up to day 169
  The incidence of Adverse Events(AEs)and Serious Adverse Events(SAEs)from treatment until the last scheduled follow-up visit
Number of subjects with abnormal vital signs | up to day 169
  Vital signs measurements will include pulse rate, respiration rate, blood pressure (systolic and diastolic blood pressure) and body temperature.
Number of subjects with abnormal clinically significant results from physical examination | up to day 169
  The physical examinations will include examination of the following: skin and mucous membranes, lymph nodes, head and neck, chest, abdomen, musculoskeletal, nervous system, and other sites of note elicited from the subject.
Number of subjects with abnormal clinically significant 12-lead electrocardiogram (ECG) parameters | up to day 169
  The examination indicators include heart rate, PR, QRS, uncorrected QT, and QTcF(corrected by Fridericia formula).
Number of subjects with abnormal clinically significant clinical laboratory results | up to day 169
  Clinical laboratory tests include hematology, urinalysis, blood chemistry, coagulation function.

SECONDARY OUTCOMES:
Concentration of 9MW3011 in serum | up to day 169
PD-parameters-hepcidin | up to day 169
  Change from baseline in hepcidin levels
PD-parameters-serum iron | up to day 169
  Change from baseline in serum iron levels
Anti-drug antibody(ADA) | up to day 169
  The incidence of ADA
Liver iron concentration(LIC) | up to day 169
  Change from baseline in LIC

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The first Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No